CLINICAL TRIAL: NCT03940066
Title: Evaluation of Ambulatory Monitoring of Patients After High-risk Acute Coronary Syndrome Using Two Different Systems: Biomonitor-2 and Kardia Mobile
Acronym: Monitor- ACS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación EPIC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Monitor- ACS - EPIC 013
Record Dates: First submitted 2019-05-05; First posted 2019-05-07 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2023-04

CONDITIONS: Atrial Fibrillation; Syncope; Tachycardia; Arrhythmias, Cardiac; Heart Diseases
Keywords: Cardiac Monitor
MeSH Terms: conditions — Atrial Fibrillation; Syncope; Tachycardia; Arrhythmias, Cardiac; Heart Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Monitoring group (Other)
  Interventions: Device: Biomonitor-2 and Kardia mobile
- Standard Care (Other)
  Interventions: Other: No Intervention

INTERVENTIONS:
Device: Biomonitor-2 and Kardia mobile — Implantable cardiac monitor and Smart-phone based electrocardiogram recording
  Arms: Monitoring group
Other: No Intervention — No intervention
  Arms: Standard Care

SUMMARY:
The objective of the study is to evaluate the efficacy of monitoring after discharge of patients with high-risk acute coronary syndrome.

DETAILED DESCRIPTION:
The objective of the study is to evaluate the efficacy of monitoring after discharge of patients with high-risk acute coronary syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Patient is able to understand the nature of study and has provided written informed consent.
* Patient with Acute Coronary Syndrome, with or without elevation of the ST segment at the EKG (the last with elevation of troponins).
* Patient with coronariography at the episode of ACS showing severe lesions treated with stent.
* Patient with risk index for 6-month mortality (GRACE score) of more than 118.
* Patient with risk index for stroke (CHA2DS2-VACS score) of more than 2.

Exclusion Criteria:

* Patient with history of AF.
* Patient with episodes of AF during admission at the current episode.
* Patient with pacemaker or ICD (implantable cardioverter-defibrillator) previously.
* Patient with indication of pacemaker or ICD in current or short-term phase.
* Patient is participating in another interventional clinical investigation.
* Patient is pregnant or breast feeding.
* Patient´s life-expectancy is less than 24 months.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2019-11-12 (Actual); Primary Completion 2024-04-08 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Atrial fibrilation (AF / atrial flutter) | 1 year
  Detection rates for atrial fibrilation (AF / atrial flutter) during the follow up.
Ventricular arrhythmia in the electrocardiogram (EKG) | 1 year
  Detection rates of ventricular arrhythmia in the electrocardiogram (EKG) during the follow up.
Advanced conduction abnormalities and significant ST shifts (> 1 mm) in the EKG | 1 year
  Detection rates of advanced conduction abnormalities and significant ST shifts (> 1 mm) in the EKG.

SECONDARY OUTCOMES:
Major Adverse Cardiovascular and Cerebrovascular Events (MACCE) | 1 year
  MACCE rates defined as cardiovascular and cerebrovascular events during the follow up.
Re-hospitalization | 1 year
  Number of Re-hospitalization during the follow up.
Correlation of primary outcomes between Biomonitor-2 versus Kardia Mobile | 1 year
  Correlation of primary outcomes between Biomonitor-2 versus Kardia Mobile during the follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Felipe Rodríguez Entem, MD, PhD, Principal Investigator — Hospital Universitario Marqués de Valdecilla; José M De la Torre Hernández, MD, PhD, Principal Investigator — Hospital Universitario Marqués de Valdecilla
Locations (1):
- Hospital Universitario Marques de Valdecilla, Santander, Spain

REFERENCES:
- [Background] Jernberg T, Hasvold P, Henriksson M, Hjelm H, Thuresson M, Janzon M. Cardiovascular risk in post-myocardial infarction patients: nationwide real world data demonstrate the importance of a long-term perspective. Eur Heart J. 2015 May 14;36(19):1163-70. doi: 10.1093/eurheartj/ehu505. Epub 2015 Jan 13. PMID 25586123
- [Background] Bhatt DL, Eagle KA, Ohman EM, Hirsch AT, Goto S, Mahoney EM, Wilson PW, Alberts MJ, D'Agostino R, Liau CS, Mas JL, Rother J, Smith SC Jr, Salette G, Contant CF, Massaro JM, Steg PG; REACH Registry Investigators. Comparative determinants of 4-year cardiovascular event rates in stable outpatients at risk of or with atherothrombosis. JAMA. 2010 Sep 22;304(12):1350-7. doi: 10.1001/jama.2010.1322. Epub 2010 Aug 30. PMID 20805624
- [Background] Eagle KA, Lim MJ, Dabbous OH, Pieper KS, Goldberg RJ, Van de Werf F, Goodman SG, Granger CB, Steg PG, Gore JM, Budaj A, Avezum A, Flather MD, Fox KA; GRACE Investigators. A validated prediction model for all forms of acute coronary syndrome: estimating the risk of 6-month postdischarge death in an international registry. JAMA. 2004 Jun 9;291(22):2727-33. doi: 10.1001/jama.291.22.2727. PMID 15187054
- [Background] Chua SK, Lo HM, Chiu CZ, Shyu KG. Use of CHADS(2) and CHA(2)DS(2)-VASc scores to predict subsequent myocardial infarction, stroke, and death in patients with acute coronary syndrome: data from Taiwan acute coronary syndrome full spectrum registry. PLoS One. 2014 Oct 24;9(10):e111167. doi: 10.1371/journal.pone.0111167. eCollection 2014. PMID 25343586
- [Background] Halcox JPJ, Wareham K. Response by Halcox and Wareham to Letter Regarding Article, "Assessment of Remote Heart Rhythm Sampling Using the AliveCor Heart Monitor to Screen for Atrial Fibrillation: The REHEARSE-AF Study". Circulation. 2018 May 15;137(20):2193-2194. doi: 10.1161/CIRCULATIONAHA.118.033773. No abstract available. PMID 29760234
- [Derived] De La Torre Hernandez JM, Exposito V, Gonzalez Enriquez S, Rodriguez Entem F, Margarida A, Garcia Camarero T, Veiga G, Sainz Laso F, Lee DH, Gil Ongay A, Barrera S, Catoya S, Garilleti C, Hernandez R, Obregon C, Olalla JJ. Evaluation of ambulatory electrocardiographic monitoring of patients after high-risk acute coronary syndrome: the MONITOR ACS-Epic 13 randomized trial. Front Cardiovasc Med. 2025 Aug 18;12:1646175. doi: 10.3389/fcvm.2025.1646175. eCollection 2025. PMID 40901364